CLINICAL TRIAL: NCT01874899
Title: Prospective Randomized Feasibility Study Comparing Manual vs. Automatic Position-Adaptive Spinal Cord Stimulation With Surgical Leads
Acronym: RestoreSensor
Status: Completed | Type: Observational
Sponsor: Justin Parker Neurological Institute (Other)
Responsible Party: Principal Investigator, Alan T. Villavicencio, MD, Principle Investigator, Justin Parker Neurological Institute
Other Study IDs: JPNI-3
Record Dates: First submitted 2013-06-06; First posted 2013-06-11 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Chronic Refractory Low Back and Leg Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Manual, then Automatic Stimulation: The RestoreSensor neurostimulator will be programed for manual stimulation adjustments and the patients will crossover to automatic stimulation group after 1.5 months
  Interventions: Device: RestoreSensor Neurostimulation
- Automatic, then Manual Stimulation: The RestoreSensor neurostimulator will be programed for automatic stimulation adjustments and the patients will crossover to manual stimulation group after 1.5 months.
  Interventions: Device: RestoreSensor Neurostimulation

INTERVENTIONS:
Device: RestoreSensor Neurostimulation

SUMMARY:
The main purpose of this study is to establish the extent that chronic pain patients implanted with surgical, laminectomy-type, leads experience position-related variation in spinal cord stimulation therapy and to investigate the effects of manual versus automatic position-adaptive spinal cord stimulation on clinical outcome.

DETAILED DESCRIPTION:
A single-center, prospective, randomized study with a two-arm crossover design. The primary objective of this study is to establish threshold and therapeutic stimulation parameters for the RestoreSensor neurostimulator in response to postural changes. The secondary objective is to compare the effectiveness of spinal cord stimulation with manual versus automatic position-adaptive settings for chronic refractory low back and/or extremity pain.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature adults between 18 and 70 years old
* Patients with chronic refractory back and/or leg pain associated with failed back surgery syndrome, post-laminectomy pain, radicular pain syndrome or radiculopathy refractory to conservative and surgical interventions
* > 50% pain reduction during the trail period
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing to sign a study specific informed consent

Exclusion Criteria:

* Previous SCS treatment
* Surgically remediable spinal condition
* Active local or systemic infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic refractory back and leg pain associated with failed back surgery syndrome, post-laminectomy pain, radicular pain syndrome or radiculopathy refractory to conservative and surgical interventions.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Stimulation amplitude changes in response to postural changes | 6 months
  Threshold and therapeutic stimulation parameters in different postures: lying right, lying left, lying prone, lying supine, upright and upright active will be collected for manual and sensor-driven position-adaptive stimulation.

SECONDARY OUTCOMES:
Sleep quality improvement | 6 months
  Pittsburg Sleep Quality Index Oswestry Disability Index

OTHER OUTCOMES:
Disability score improvement | 6 months
  Oswestry Disability Index
Pain scores | 6 months
  Numeric pain scale
Patient satisfaction | 6 months
  Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Kara Beasley, DO, Principal Investigator — Boulder Neurosurgical Associates
Locations (1):
- Boulder Neurosurgical Associates, Boulder, Colorado, United States